CLINICAL TRIAL: NCT05518448
Title: The Effect of a Ketone Drink on Liver Glucose Production in People With Type 2 Diabetes
Acronym: KES2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 22-02-02-B-01
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus; Ketosis
Keywords: Diabetes; Exogenous ketones; Postprandial glycemia; Endogenous glucose production
MeSH Terms: conditions — Diabetes Mellitus; Ketosis

STUDY DESIGN:
Intervention Model Description: Ketone vs placebo crossover
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone (Experimental): Ketone monester (beta-hydroxybutyrate (β-OHB)
  Interventions: Dietary Supplement: Ketone - beta-hydroxybutyrate (β-OHB)
- Placebo (Placebo Comparator): Non-caloric placebo
  Interventions: Dietary Supplement: Ketone - beta-hydroxybutyrate (β-OHB)

INTERVENTIONS:
Dietary Supplement: Ketone - beta-hydroxybutyrate (β-OHB) — Ketone - beta-hydroxybutyrate (β-OHB)

SUMMARY:
What is the effect of a ketone drink on liver glucose production, and postprandial glycemia, in people with type 2 diabetes.

DETAILED DESCRIPTION:
Background: Ketones are molecules that are naturally produced by our body during fasting or diets low in carbohydrates. Ketones can affect how our liver produces and maintains our body's blood sugar levels, which could be important in the management of type 2 diabetes (T2D), where high blood sugar levels are partly because of excess sugar production by the liver.

Objectives: To determine if, and how, a ketone drink can lower blood glucose in people with T2D following a meal.

Methods: Twelve people with T2D will visit our laboratory in the morning on two occasions and ingest a drink containing ketones or placebo on each visit in a random order before ingesting a milkshake style drink containing sugar. Blood samples will then be taken at regular intervals over 4 hours to determine if the ketone drink has lowered blood sugar levels in response to the meal, and if this was due to reduced sugar production by the liver.

Value: This research will provide new knowledge about the regulation of liver blood sugar production in response to ketone ingestion. This may also inform future clinical trials to establish if ketone drinks could be used as a treatment for T2D.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes by a physician, a current HbA1c of 6.5-8.5%, and receiving treatment with lifestyle advice or oral glucose-lowering medications.
* Non-smoking
* Blood pressure <160/100 mm/Hg

Exclusion Criteria:

* Exogenous insulin or SGLT2 inhibitors for type 2 diabetes treatment.
* Following a low-carbohydrate ketogenic diet, periodic fasting diet, or consuming ketogenic supplements.
* Other diagnosed chronic metabolic, cardiovascular, respiratory, neurological, or gastrointestinal disease.
* Smoker
* Blood pressure >160/100 mm/Hg
* Lactose intolerant

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
EGP | 6 hours
  Endogenous glucose production

SECONDARY OUTCOMES:
Postprandial glycemia | 4 hours
  Postprandial glucose concentrations
Insulin | 6 hours
  Serum insulin concentration
Plasma β-OHB | 6 hours
  Plasma β-OHB concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- Sport & Health Sciences, University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Monteyne AJ, Falkenhain K, Whelehan G, Neudorf H, Abdelrahman DR, Murton AJ, Wall BT, Stephens FB, Little JP. A ketone monoester drink reduces postprandial blood glucose concentrations in adults with type 2 diabetes: a randomised controlled trial. Diabetologia. 2024 Jun;67(6):1107-1113. doi: 10.1007/s00125-024-06122-7. Epub 2024 Mar 14. PMID 38483543